CLINICAL TRIAL: NCT02235454
Title: A Prospective Evaluation of the Novel Glaucoma Premium Edition Software for Spectral Domain Optical Coherence Tomography
Brief Title: SDOCT-GMPE Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00056471
Record Dates: First submitted 2014-09-05; First posted 2014-09-10 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Glaucoma
Keywords: glaucoma; OCT; spectral domain optical coherence tomography
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glaucoma arm (Other): Consecutive patients with glaucoma will undergo non-invasive OCT imaging
  Interventions: Device: SDOCT-GMPE software

INTERVENTIONS:
Device: SDOCT-GMPE software — Noninvasive imaging of the optic nerve in patients with existing glaucoma

SUMMARY:
The investigators prospectively evaluate the new glaucoma premium edition (GMPE) software for spectral domain optical coherence tomography (SDOCT) and if this software is superior to the conventional one that is currently used for SDOCT.

DETAILED DESCRIPTION:
The new GMPE software can now identify the ocular structures without input from the operator thus reducing operator induced errors. It also measures the thickness of the entire optic nerve head so as to allow for another anatomic area of the eye to be measured for assessment of glaucoma. In addition, it permits collection of retinal nerve fiber layer thickness data in three concentric circles instead of just one in order to account for different sizes of optic nerves.

Subjects who are receiving routine SDOCT (CPT 92133) will be recruited from the Duke Eye Center and its associated satellite clinics. Following informed consent, subjects undergo additional imaging using the SDOCT-GMPE software at the Duke Eye Center and its associated satellite clinics. The imaging results may be used in clinical care for the subjects.

ELIGIBILITY:
Inclusion Criteria:

* capable and willing to provide consent
* history of clinically-diagnosed glaucoma
* at least 18 years of age

Exclusion Criteria:

* unable or unwilling to give consent
* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Asrani, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glaucoma Arm
Started | 57
Completed | 55
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Glaucoma Arm
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 39
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Retinal Nerve Fiber Layer (RNFL) Thickness Correlation Width Global Bruch's Membrane Opening-minimum Rim Width (BMO-MRW)
Description: Pearson correlation coefficient between Retinal Nerve Fiber Layer (RNFL) thickness correlation width global Bruch's membrane opening-minimum rim width (BMO-MRW).
Time Frame: imaging approximately 10 minutes
Population: All usable images of one eye of each participant
Measure: Number; unit: correlation coefficient
Arm/Group | Glaucoma Arm
Number analyzed (Participants) | 49
correlation coefficient | 0.70

ADVERSE EVENTS:
Time Frame: During measurement time (approximately ten minutes)
Groups:
- Glaucoma Arm: Consecutive willing patients with glaucoma will undergo non-invasive OCT imaging
  SDOCT-GMPE software: Noninvasive imaging of the optic nerve in patients with existing glaucoma
Arm/Group | Glaucoma Arm
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes